CLINICAL TRIAL: NCT05174598
Title: A Phase III, Multicentre, Randomized, Observer Blind, Parallel Group, Three Arms, Controlled Clinical Trial to Evaluate the Efficacy and Safety of Topically Applied Calcipotriol/AKVANO 50 μg/g Cutaneous Solution Against Calcipotriol Ointment 50 Micrograms/g, Sandoz and Placebo in Patients With Mild to Moderate Plaque Psoriasis
Brief Title: A Clinical Trial to Evaluate Efficacy and Safety of Two Different Formulations of Topical Calcipotriol in Patients With Mild to Moderate Plaque Psoriasis
Acronym: AKP01
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cadila Pharnmaceuticals (Industry)
Collaborators: Lipidor AB, Svärdvägen 13 SE-182 33 Danderyd, Sweden (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRSC16004
Record Dates: First submitted 2021-11-30; First posted 2022-01-03 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: Mild to Moderate Plaque Psoriasis
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Calcipotriol/AKVANO, 50 μg/g cutaneous solution (Experimental): Spray formulation applied topically, twice daily, for the duration of 8 weeks.
  Interventions: Drug: Calcipotriol/AKVANO, 50 μg/g cutaneous solution
- Calcipotriol Ointment 50 micrograms/g, Sandoz (Active Comparator): Ointment applied topically, twice daily, for the duration of 8 weeks.
  Interventions: Drug: Calcipotriol Ointment 50 micrograms/g
- Placebo (Placebo Comparator): Spray formulation applied topically, twice daily, for the duration of 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Calcipotriol/AKVANO, 50 μg/g cutaneous solution — Topical spray formulation containing Calcipotriol 50 μg/g. Twice daily treatment by spraying on a psoriasis affected area for 8 weeks.
  Arms: Calcipotriol/AKVANO, 50 μg/g cutaneous solution
Drug: Calcipotriol Ointment 50 micrograms/g — Topical Ointment formulation containing Calcipotriol 50 micrograms/g. Twice daily treatment by applying on a psoriasis affected area for 8 weeks.
  Arms: Calcipotriol Ointment 50 micrograms/g, Sandoz
Other: Placebo — Topical spray formulation containing Vehicle of test formulation. Twice daily treatment by spraying on a psoriasis affected area for 8 weeks.
  Arms: Placebo

SUMMARY:
This study is a Phase III, multicentre, randomized, observer blind, parallel group, three arms, controlled clinical trial to evaluate the efficacy and safety of topically applied Calcipotriol/AKVANO 50 μg/g cutaneous solution against Calcipotriol Ointment 50 micrograms/g, Sandoz and placebo in patients with mild to moderate plaque psoriasis

DETAILED DESCRIPTION:
Total 278 patients with mild to moderate plaque psoriasis were randomized into the study. Study medications were applied twice daily for 8 weeks of study duration.

Patient's condition was assessed using of Physician's Global Assessment (PGA) and PASI Scale.

Primary objective of this study is to assess the therapeutic equivalence of Calcipotriol/AKVANO, 50 μg/g cutaneous solution with Calcipotriol Ointment 50 micrograms/g, Sandoz based on PASI score.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients (Non-pregnant) of plaque psoriasis aged 18 to 65 years having either Fitzpatrick skin type I-III or IV-VI.<br/>
* Diagnosis of stable plaque psoriasis for 6 month by a dermatologist with lesions on arms, legs or trunk.
* Mild to moderate psoriasis on Physician's global assessment (PGA),
* Body Surface Area (BSA) involvement of 5-10% (both included) and PASI ≥ 5.
* Patients must be willing to provide written informed consent and willing to comply with study requirements

Exclusion Criteria:

* Predominantly palmo-plantar, flexural, scalp and nail location of psoriasis
* Guttate, erythrodermic, or pustular psoriasis as sole or predominant form of psoriasis.
* Patient with any uncontrolled systemic disease
* Patient with positive serology tests like HIV, HCV & HBsAg.
* Patient with presence of any skin disease that might interfere with the diagnosis or evaluation of the test medications.
* Patient with spontaneously improving or rapidly deteriorating plaque psoriasis.
* Use of systemic agents within four weeks prior to screening.
* Use of biologic agents within four weeks prior to study entry.
* Use of topical drugs that might alter the course of psoriasis or has received ultraviolet B treatment within two weeks prior to study entry.
* Use of phototherapy with psoralen ultraviolet A treatment within four weeks prior to study entry.
* Known sensitivity to any of the study treatments and/or study treatment's components.
* Need for surgery or hospitalization during the study
* Pregnant or nursing Female patient or planning a pregnancy
* Concurrent involvement in any other clinical study within 30 days prior to entering the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Change in Psoriasis Area and Severity Index | Baseline to 8 weeks Post-randomization
  Assessment of severity of psoriasis by comparing the change in Psoriasis Area and Severity Index between test and comparator (score ranging from 0 to 72, higher score means worsening of the disease)

SECONDARY OUTCOMES:
Assessment of Physician's Global Assessment (PGA) | Baseline to 2, 4 and 8 weeks of treatment Post-randomization
  Proportion of patients achieving PGA 0 or 1 with Test and comparator
Incidence of Adverse Events and SAEs (Safety and Tolerability) | Till 8 weeks Post-randomization
  Incidence of Adverse Event and Serious Adverse Event between three treatment arms
More than 50 % reduction in PASI Score (PASI 50) | Baseline to 2, 4 and 8 weeks of treatment Post-randomization
  Proportion of patients achieving >50 % reduction in PASI Score (PASI50) with Test and comparator
More than 75 % reduction in PASI Score (PASI 75) | Baseline to 2, 4 and 8 weeks of treatment Post-randomization
  Proportion of patients achieving >75 % reduction in PASI Score (PASI75) with Test and comparator.
Change in Irritation based on Visual Analogue scale (VAS) | Baseline to 2, 4 and 8 weeks of treatment Post-randomization
  To evaluate change in irritation based on Visual Analogue scale between three treatment arms Visual Analogue scale (VAS) ranges from 0 to 10 (higher scores mean worse outcome)
Change in itching based on Visual Analogue scale | Baseline to 2, 4 and 8 weeks of treatment Post-randomization
  To evaluate change in itching based on Visual Analogue scale between three treatment arms, Visual Analogue scale (VAS) ranges from 0 to 10 (higher scores mean worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Avhad, MBBS, Study Director — Cadila Pharmaceuticals Limited
Locations (14):
- India (14):
  - AC Subbareddy Government Hospital, Nellore, Andhra Pradesh
  - Downtown Hospital, Guwahati, Assam
  - Marwari Hospital & Research Centre, Guwahati, Assam
  - Sanjeevani CBCC USA Cancer Hospital, Raipur, Chhattisgarh
  - Kanoria Hospital & Research Centre, Gandhinagar, Gujarat
  - GMERS Medical College & Hospital, Vadodara, Gujarat
  - Dhiraj General Hospital, Vadodara, Gujarat
  - KLES Dr. Prabhakar Kore Hospital & Medical Reserach Centre, Belagavi, Karnataka
  - Government Medical College, Aurangabad, Maharashtra
  - Gokuldas Tejpal Hospital Grant Government Medical College & Sir JJ Group of Hospital, Mumbai, Maharashtra
  - Dr. D.Y. Patil Hospital, Mumbai, Maharashtra
  - Midland Healthcare & Research Center, Lucknow, Uttar Pradesh
  - Surya Super Speciality Hospital, Varanasi, Uttar Pradesh
  - Postgraduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: No